CLINICAL TRIAL: NCT07379411
Title: Energy-based Opportunistic Salpingo-oophorectomy During Vaginal Hysterectomy - is it Better Than Conventional "Knot-and-cut" Approach? A Randomized Controlled Study
Brief Title: Are There Benefits of Using Energy-based Devices for Opportunistic Salpingo-oophorectomy During Vaginal Hysterectomy Compared to a Standard Cold Approach?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Michael Babin, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0119-24-WOMC
Record Dates: First submitted 2026-01-06; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: pelvic organ prolapse; vaginal surgery; vaginal hysterectomy; salpingo-oophorectomy; prophylactic salpingo-oophorectomy; vaginal salpingo-oophorectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Technique group (Active Comparator): Salpingo-oophorectomy performed using the standard surgical technique of clamping, cutting, and suturing during vaginal hysterectomy.
  Interventions: Procedure: Standard salpingo-oophorectomy technique
- LigaSure Maryland group (Experimental): Salpingo-oophorectomy performed using the LigaSure Maryland energy-based vessel sealing device during vaginal hysterectomy
  Interventions: Device: LigaSure MaryLand

INTERVENTIONS:
Device: LigaSure MaryLand — Energy-based vessel sealing device used to perform salpingo-oophorectomy.
  Arms: LigaSure Maryland group
Procedure: Standard salpingo-oophorectomy technique — Salpingo-oophorectomy performed using clamping, cutting, and suturing without the use of energy-based devices.
  Arms: Standard Technique group

SUMMARY:
This study compares two methods for removing the fallopian tubes and ovaries during vaginal hysterectomy for pelvic organ prolapse.

One method uses an energy-based surgical device called LigaSure Maryland, which seals blood vessels using electrical energy. The other method is the standard surgical approach, which involves clamping, cutting, and suturing the tissue. The purpose of the study is to determine whether the use of the LigaSure device is as safe as, or more effective than, the standard technique, in terms of procedure duration, blood loss, postoperative pain, length of hospital stay, and complication rates.

Women who are scheduled to undergo vaginal hysterectomy for pelvic organ prolapse and for whom removal of the fallopian tubes and ovaries is recommended may participate in the study. Participants will be randomly assigned to one of two groups, receiving either the LigaSure technique or the standard surgical technique.

The decision to perform removal of the fallopian tubes and ovaries will be made before surgery based on standard medical indications. Participants will not be informed which surgical technique is used during their operation. Surgical outcomes between the two groups will be compared to evaluate safety and effectiveness.

DETAILED DESCRIPTION:
Vaginal hysterectomy is a common surgical procedure performed for benign gynecologic indications, including pelvic organ prolapse. Opportunistic salpingectomy, with or without oophorectomy, is increasingly recommended at the time of hysterectomy in women at average risk for ovarian cancer, as it may reduce future cancer risk without increasing surgical morbidity. During vaginal hysterectomy, salpingo-oophorectomy can be performed using a conventional surgical technique involving clamping, cutting, and suturing, or by using energy-based vessel sealing devices.

Energy-based devices, such as the LigaSure Maryland, have been shown in other gynecologic procedures to reduce operative time, blood loss, and length of hospital stay. However, there are limited data comparing energy-based versus conventional techniques specifically for opportunistic salpingo-oophorectomy performed during vaginal hysterectomy.

This prospective, randomized controlled study is designed to compare an energy-based technique using the LigaSure Maryland device with a standard "knot-and-cut" technique for opportunistic salpingo-oophorectomy during vaginal hysterectomy for benign indications.

Women scheduled to undergo vaginal hysterectomy for pelvic organ prolapse, for whom salpingo-oophorectomy is recommended according to standard clinical indications, will be eligible for participation. After providing informed consent, participants will be randomly assigned to one of two parallel groups. In the intervention group, salpingo-oophorectomy will be performed using the LigaSure Maryland energy-based vessel sealing device. In the control group, salpingo-oophorectomy will be performed using the standard surgical technique of clamping, cutting, and suturing.

Randomization will be performed prior to surgery using a computerized randomization tool. Participants will be blinded to the surgical technique used. Surgeons will not be blinded due to the nature of the interventions.

The primary outcome of the study is the duration of the salpingo-oophorectomy procedure, measured from completion of the vaginal hysterectomy and the decision to proceed with salpingo-oophorectomy until removal of the fallopian tube and ovary specimen on both sides. Secondary outcomes include estimated blood loss during the procedure, postoperative pain assessed using a visual analog scale (VAS), length of postoperative hospital stay, and the rate of intraoperative and postoperative complications.

Both surgical techniques are considered standard of care and are commonly used in modern gynecologic surgery. Patient safety is not expected to be compromised by participation in either study group. In cases where deviation from the assigned surgical technique is required intraoperatively due to anatomical or technical considerations, the participant will be excluded from the final analysis to avoid bias.

The results of this study aim to provide evidence regarding the safety and efficacy of energy-based opportunistic salpingo-oophorectomy during vaginal hysterectomy and may help guide surgical decision-making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Scheduled to undergo vaginal hysterectomy for pelvic organ prolapse.
* Recommended to undergo opportunistic salpingo-oophorectomy according to standard clinical indications.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Suspected or known pelvic malignancy.
* Lack of informed consent.
* Planned opportunistic salpingo-oophorectomy using a non-vaginal surgical approach.
* Planned opportunistic salpingo-oophorectomy using a vNOTES (vaginal natural orifice transluminal endoscopic surgery) approach.
* Intraoperative need to deviate from the assigned surgical technique due to anatomical or technical considerations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Duration of salpingo-oophorectomy procedure | From completion of vaginal hysterectomy until completion of salpingo-oophorectomy, assessed over approximately 5-30 minutes during surgery
  Duration of the salpingo-oophorectomy procedure, measured from completion of the vaginal hysterectomy and the decision to proceed with salpingo-oophorectomy until removal of the fallopian tube and ovary specimen from the patient on the both sides.

SECONDARY OUTCOMES:
Intraoperative blood loss | From completion of vaginal hysterectomy until completion of salpingo-oophorectomy, assessed over approximately 5-30 minutes during surgery
  Blood loss during salpingo-oophorectomy, measured by weighing surgical pads used during the procedure
Postoperative pain | Within 24 hours after surgery
  Postoperative pain assessed using a visual analog scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain), as routinely used in the gynecology department, assessed at the evening of the day of surgery
Length of hospital stay | From admission to the gynecology ward after surgery until hospital discharge, assessed over approximately 1-5 days
  Duration of postoperative hospitalization measured from admission to the gynecology until discharge decision by the attending surgeon
Intraoperative and postoperative complications | From surgery to 30 days after surgery
  Rate of intraoperative and postoperative complications related to the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kahn RM, Gordhandas S, Godwin K, Stone RL, Worley MJ Jr, Lu KH, Long Roche KC. Salpingectomy for the Primary Prevention of Ovarian Cancer: A Systematic Review. JAMA Surg. 2023 Nov 1;158(11):1204-1211. doi: 10.1001/jamasurg.2023.4164. PMID 37672283
- [Result] Bonavina G, Busnelli A, Salmeri N, Cavoretto PI, Salvatore S, Candiani M, Bulfoni A. Opportunistic salpingectomy at the time of vaginal hysterectomy: A systematic review and meta-analysis. Int J Gynaecol Obstet. 2024 Aug;166(2):494-501. doi: 10.1002/ijgo.15386. Epub 2024 Jan 21. PMID 38247214
- [Result] Antosh DD, High R, Brown HW, Oliphant SS, Abed H, Philip N, Grimes CL. Feasibility of prophylactic salpingectomy during vaginal hysterectomy. Am J Obstet Gynecol. 2017 Nov;217(5):605.e1-605.e5. doi: 10.1016/j.ajog.2017.07.017. Epub 2017 Jul 20. PMID 28734829
- [Result] Kroft J, Selk A. Energy-based vessel sealing in vaginal hysterectomy: a systematic review and meta-analysis. Obstet Gynecol. 2011 Nov;118(5):1127-1136. doi: 10.1097/AOG.0b013e3182324306. PMID 22015881
- [Result] Lauterbach R, Gruenwald O, Matanes E, Justman N, Mor O, Vitner D, Avrahami R, Ghanem N, Zipori Y, Weiner Z, Lowenstein L. A randomized controlled trial of 2 techniques of salpingectomy during cesarean delivery. Am J Obstet Gynecol MFM. 2022 Nov;4(6):100690. doi: 10.1016/j.ajogmf.2022.100690. Epub 2022 Jul 16. PMID 35843545